CLINICAL TRIAL: NCT06215690
Title: Evaluation of Anterior Middle Brain Structures With Cerebrovascular Flow in Fetuses With Fetal Growth Restriction
Status: Active, not recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Can Ozan Ulusoy, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: AEŞH-EK1-2023-066
Record Dates: First submitted 2023-12-22; First posted 2024-01-22 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Fetal Growth Retardation; Fetal Neurodevelopmental Disorder
Keywords: Fetal Growth Restriction; Anterior Middle Brain Structures; Cerebrovascular Flow
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Women with Fetal Growth Restriction: Fetuses with fetal growth restriction according to Delphi consensus criteria between 32-37 weeks of gestation
  Interventions: Diagnostic Test: Ultrasound measurements
- Healthy Pregnancies: Normally developing fetuses between 32-37 weeks of gestation
  Interventions: Diagnostic Test: Ultrasound measurements

INTERVENTIONS:
Diagnostic Test: Ultrasound measurements — Evaluation will be performed by ultrasonography. The following measurements will be taken with the ultrasonographic examination.
  * BPD (Biparietal Diameter)
  * HC (Head Circumference)
  * AC (Abdominal Circumference)
  * FL (Femur Length)
  * EFW (Estimated Fetal Weight)
  * Umbilical Artery Doppler Sistole/Diastole (S/D) ,Pulsatility İndex (PI), Resistance İndex (RI)
  * Middle Cerebral Artery S/D,PI,RI
  * Uterine Artery Doppler PI
  * Anterior Cerebral Artery S/D,PI,RI
  * CPUR (Cerebral - Placental - Uterin PI Ratio)
  * CPR (Cerebral - Placental PI Ratio)
  * The deepest free single vertical pocket in the amnion mai
  * Cavum Septum Pellucidum: Width - Length Diameters
  * OFD (Occipitofrontal length)
  * FAPD (Frontal Anterior Posterior Diameter)
  * FAPD/OFD ratio
  * Cerebellar diameter
  * Lateral ventricle depth
  * Insular depth
  * Sylvian fissure depth

SUMMARY:
The study will be conducted to examine the effects of abnormal growth pattern and cerebrovascular blood flow measurements on fetal frontal lobe development with the advancing ultrasound technology. Antenatal assessment of frontal lobe development will enable clinicians to predict neurodevelopmental problems that may develop postnatally. In addition, this study will examine the effects of FGR on frontal lobe development.

DETAILED DESCRIPTION:
Fetal growth restriction (FGR) affects up to 10% of all pregnancies. The International Society of Ultrasound in Obstetrics & Gynecology (ISUOG) adopts the Delphi consensus criteria for the definition of FGR. These criteria include estimated fetal weight (EFW) or abdominal circumference (AC) < 3rd percentile or EFW or AC < 10th percentile with abnormal Doppler findings or decreased growth percentiles. FGR is a cause of perinatal morbidity and mortality. These perinatal outcomes include cardiovascular, endocrine and neurodevelopmental disorders. Fetal growth restriction, which is associated with lower neurobehavioral test scores, is associated with significant postnatal costs for both the health care system and families. Previous literature has shown that three-dimensional ultrasonography of intracranial structures reveals significant differences between fetuses with FGR and gestational age-appropriate (AGA) fetuses. However, the limited use of three-dimensional ultrasonography has hindered clinical applications. The frontal Anterior-Posterior Diameter (FAPD)/Occipital-Frontal Diameter (OFD) ratio has recently been used to assess frontal lobe development in fetuses with congenital heart disease. The FAPD is obtained by measuring from the inner line of the frontal bone along the fetal brain midline to the posterior edge of the CSP. This measurement refers to the frontal lobe of the fetal cerebrum. This study was designed to investigate the FAPD/ OFD ratio and frontal lobe development in fetuses with FGR and to evaluate cerebrovascular flow and anterior midbrain structures in FGR fetuses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy hearts between the ages of 18-40
* Singleton pregnancies
* 32 to 37 weeks gestational week range

Exclusion Criteria:

* Multiple pregnancies
* Fetuses with fetal karyotype abnormalities
* Pregnant women with co-morbidity
* Fetuses with fetal intracranial hemorrhage
* Fetuses with cranial anomalies
* Maternal obesity preventing measurement

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will include normally developing fetuses between 32-37 weeks of gestation and fetuses with fetal growth restriction.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-07-04 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
Ultrasonographic measurements and comparison of fetuses with and without fetal growth retardation | Prenatal (32-37 gestational weeks)
  Demographic data, ultrasonographically obtained biometric measurements, and Doppler flow data will be compared in both groups.
  * Frontal Anterior Posterior Length, Occipital to Frontal Diameter ratio mm/mm (FAPD mm/OFD mm)
  * Cerebellar length, head circumference length ratio mm/mm (CD mm / HC mm)
  The main biometric measurement of the study will be comparison.
  The percentile values of the Anterior Cerebral Artery Doppler Pulsatility Index (cm/s) (ACA PI cm/s ) and Middle Cerebral Artery Doppler Pulsatility Index cm/s (MCA PI cm/s) will be calculated for the week of ultrasonographic measurement, and the ratio of ACA PI and MCA PI will be compared in fetuses with and without fetal growth retardation.

SECONDARY OUTCOMES:
Evaluation of neonatal findings of the patients included in the study | through study completion, an average of 4 months
  Fetuses included in the study will be evaluated after delivery.
  Whether there is a need for Neonatal Intensive Care, APGAR scores, (0-10) Whether neonatal complications develop,
  will be evaluated and compared in the control group and in the group with fetal growth retardation.

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In accordance with hospital policy, it is not allowed to share data with third parties. If necessary, the chief researcher can be contacted

REFERENCES:
- [Derived] Ulusoy CO, Agaoglu RT, Sucu ST, Kurt DS, Bucak M, Seyhanli Z, Yucel KY. Evaluation of Anterior and Middle Brain Structures With Cerebrovascular Flow in Fetuses With Fetal Growth Restriction: A Prospective Study. J Clin Ultrasound. 2025 Feb;53(2):262-270. doi: 10.1002/jcu.23857. Epub 2024 Oct 8. PMID 39377442